CLINICAL TRIAL: NCT06090669
Title: Phase Ib Study of Imatinib to Increase RUNX1 Activity in Participants With Germline RUNX1 Deficiency
Brief Title: Imatinib to Increase RUNX1 Activity in Participants With Germline RUNX1 Deficiency
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001542; 001542-C
Record Dates: First submitted 2023-10-17; First posted 2023-10-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09-24

CONDITIONS: Inherited Bone Marrow Failure Syndrome; Familial Platelet Disorder With Predisposition to Myeloid Malignancies
Keywords: predisposition to hematologic malignancies; germline mutations; IBMFS
MeSH Terms: conditions — Congenital Bone Marrow Failure Syndromes | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Escalating doses of imatinib to determine the MTD
  Interventions: Drug: imatinib; Device: TruSight Oncology
- Dose Expansion (Experimental): Imatinib at the MTD
  Interventions: Drug: imatinib; Device: TruSight Oncology
- No Treatment (No Intervention): Collection of blood or marrow only. No treatment.

INTERVENTIONS:
Drug: imatinib — Imatinib at 300-400 mg PO QD based on arm assignment/dose level
  Arms: Dose Escalation; Dose Expansion
Device: TruSight Oncology — Assay sequencing platform to identify pathogenic genetic mutations in DNA and RNA
  Arms: Dose Escalation; Dose Expansion

SUMMARY:
Background:

Runt-related transcription factor 1 (RUNX1) gene regulates the formation of blood cells. People with mutations of this gene may bleed or bruise easily; they are also at higher risk of getting cancers of the blood, bone marrow, and lymph nodes.

Objective:

The purpose of the study includes determining which dose of imatinib is best for people with pathogenic or likely pathogenic RUNX1 mutations without blood cancers, and to determine whether there are any changes in platelet function and inflammatory markers.

Eligibility:

Adults aged 18 and older with RUNX1 mutations. Healthy people without this mutation, including family members of affected participants, are also needed.

Design:

Participants with the RUNX1 mutation will be screened. They will have a physical exam with blood tests. They will have a test of their heart function. They may need a new bone marrow biopsy if they haven't had one in the past year.

Imatinib is a tablet taken by mouth once a day, every day, at home. Affected participants in different parts of the study will take imatinib for either 28 days or up to 84 days. They will fill out questionnaires about how they are feeling.

For the first part of the study, participants will have blood tests every 2 weeks, either at home or at the NIH, while they are taking the imatinib. They will have a follow up visit, at home or at the NIH, when they are done taking imatinib on Day 28.

Participants on the second part of the study will come to NIH on days 1 and days 84. They will have blood tests every 2 weeks (at home or the NIH) while they are taking imatinib. They may opt to have a bone marrow biopsy repeated after they finish their course of imatinib.

Participants will have a follow-up visit (at home or the NIH) 30 days after they stop taking imatinib.

Participants who do not have the RUNX1 mutation will have 1 clinic visit. They will have blood tests. They will fill out questionnaires. They may opt to have a bone marrow biopsy.

DETAILED DESCRIPTION:
Background:

* Runt-related transcription factor 1 (RUNX1) gene is located on chromosome 21 and encodes an important regulator of hematopoiesis. People normally inherit one functional copy from each parent.
* RUNX1 function is highly dose dependent as both too little as well as too much RUNX1 activity is associated with development of hematologic malignancy. The focus of this protocol is participants with germline RUNX1 mutations resulting in too little RUNX1 activity.
* Germline heterozygous RUNX1 mutations are inherited in an autosomal dominant manner and cause a disorder called Familial Platelet Disorder with associated Myeloid Malignancy (FPDMM). Patients with one deleterious germline RUNX1 mutation often have haploinsufficiency although some mutations are associated with a dominant negative effect.
* Clinically, patients with germline RUNX1 mutations have aberrant megakaryocytic development, which often results in quantitative and/or qualitative platelet defects. Patients often have easy bleeding or bruising, although some cases are subclinical, and they may present to clinicians with hematologic malignancy.
* Patients with germline RUNX1 mutations have 35-45% lifetime risk of developing myeloid hematologic malignancies including MDS and AML. Increased risk of B-ALL, T-ALL and other hematologic malignancies is also associated with deleterious germline RUNX1 mutations.
* Deleterious RUNX1 mutations are known to be associated with high-risk malignancy with poor response to upfront chemotherapy and require hematopoietic stem cell transplantation (HSCT).
* Imatinib is a dual SFK and ABL inhibitor that is FDA approved and indicated for treatment of CML, ALL, MDS/MPD, aggressive systemic mastocytosis (ASM) as well as hypereosinophilic syndrome (HES) and chronic eosinophilic leukemia (CEL).
* ABL physically associates with RUNX1, phosphorylates key tyrosines within the RUNX1 inhibitory domain and negatively regulates RUNX1 transcriptional activity.
* We hypothesize that imatinib will decrease RUNX1 tyrosine phosphorylation thereby increasing RUNX1 protein activity to a level closer to that expected for 2 normal copies of RUNX1. We also hypothesize that normal levels of RUNX1 protein activity will ameliorate platelet dysfunction and bleeding symptoms via objective measures.
* We expect this study to inform the biologically relevant endpoints for a subsequent phase II efficacy study, which would also seek to determine if longer term imatinib administration could prevent malignant transformation.

Objectives:

* To determine the dose of imatinib for dose expansion in participants with pathogenic or likely pathogenic germline RUNX1 mutations during the dose escalation phase
* To determine the safety of imatinib in participants with pathogenic or likely pathogenic germline RUNX1 mutations during the dose expansion phase

Eligibility:

* Age >=18 years
* Participants with deleterious germline RUNX1 mutations as defined by ClinGen with adequate organ function and no history of hematologic malignancy.

Design:

* This is a phase Ib study with 2 cohorts (participants with and without pathogenic or likely pathogenic RUNX1 mutations) and 3 arms (2 for imatinib administration and 1 for biobanking control).
* A standard 3+3 non-randomized dose-escalation design will be used in the first arm, with orally administered imatinib tested at 2 dose levels from 300 to 400 mg daily for 28 days for participants with pathogenic or likely pathogenic germline RUNX1 mutations.
* Participants will have PK/PD evaluations during Arm 2 (expansion phase).
* An expansion cohort will be treated at the maximum tolerated dose (MTD) in Arm 2, daily for 12 weeks. Participants who are treated on the dose escalation phase may also be treated in the expansion phase after an appropriate wash out period of 28 days.
* The third arm is for unaffected family control participants with wildtype RUNX1 or healthy volunteers who may choose to enroll to donate blood or marrow but will not be treated.
* Up to 13 evaluable participants will be enrolled for dose escalation, 12 participants in the expansion cohort, and up to 25 unaffected controls contemporaneously whenever feasible.

ELIGIBILITY:
* INCLUSION CRITERIA- AFFECTED PARTICIPANTS ONLY
* Affected participants must have a confirmed pathogenic or likely pathogenic germline RUNX1 variant by history. ClinGen expert variant curation panel criteria for pathogenicity will be utilized.
* Affected participants must have a history of clinically significant bleeding as defined by history of abnormal ISTH-BAT score, use of anti-bleeding medications (e.g., amicar), history of platelet transfusion, abnormal PFA screen, abnormal TEG, abnormal platelet aggregation or abnormal platelet electron microscopy.
* Bone marrow morphology, flow cytometry and cytogenetics confirmed by the NIH Department of Laboratory Medicine (DLM) at least within 12 months of initiating imatinib.
* TSO500 performed by NCI Lab of Pathology within 12 months of initiating imatinib.
* Substantial GI malabsorption is not suspected.
* Participants with human immunodeficiency virus (HIV) on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial if their HAART medications do not interact with imatinib.
* Participants with evidence of chronic hepatitis B virus (HBV) infection, on suppressive therapy with undetectable HBV viral load are eligible for this trial. Suppressive therapy medication may not interact with imatinib.
* Participants with a distant history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with active HCV infection who are currently on treatment, with undetectable HCV viral load are eligible. If unknown HCV is detected upon screening- these participants will not be eligible for the study.

INCLUSION CRITERIA- UNAFFECTED PARTICIPANTS ONLY

* Unaffected family members or healthy volunteers without RUNX1 mutation by pedigree or molecular testing Only participants who are related to the proband need to provide a molecular test.
* The last dosage of any platelet inhibiting medications was at least 2 weeks prior to enrollment and research sample acquisition.

INCLUSION CRITERIA- ALL PARTICIPANTS

* Age >=18 years.
* ECOG performance status <=2 (Karnofsky >=60%).
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes >= 3,000/mcL
  * absolute neutrophil count >= 1,500/mcL
  * platelets >= 65,000/mcL (without transfusion support)
  * total bilirubin within normal institutional limits or <= 3 X the institutional upper limit of normal for participants with Gilbert s syndrome
  * AST(SGOT)/ALT(SGPT) <= 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal.

    * NIDDK CKD-EPI equation GFR = 141 x min (Scr /kappa, 1)^alpha x max(Scr /kappa, 1)^-1.209 x 0.993^Age x 1.018 [if female] x 1.159 [if black] where: Scr is serum creatinine in mg/dL, kappa is 0.7 for females and 0.9 for males, alpha is -0.329 for females and -0.411 for males, min indicates the minimum of Scr /kappa or 1, and max indicates the maximum of Scr /kappa or 1.
    * Note: GFR is expressed in mL/min per 1.73 m^2, Scr is serum creatinine expressed in mg/dL, age is expressed in years, kappa is 0.7 for females and 0.9 for males, alpha is -0.329 for females and -0.411 for males, min indicates the minimum of Scr /kappa or 1, and max indicates the maximum of Scr /kappa or 1. Race is self-identified.
* Women of child-bearing potential and men must agree to use effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 30 days after the last administration of study drug.
* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 30 days after the last administration of study drug
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA- ALL PARTICIPANTS

* Participants who are receiving any other investigational agents.
* Participants who received prior hematologic malignancy directed therapy
* Participants receiving medication that would affect platelet number or function (e.g., aspirin and anti-platelet medications
* Participants without access to medical care at home.
* Pregnancy (confirmed with beta-HCG serum or urine pregnancy test performed in females of childbearing potential at screening).

EXCLUSION CRITERIA- AFFECTED PARTICIPANTS ONLY

* Participants with the following pathogenic/likely pathogenic abl mutations on baseline Illumina TSO500 testing of any detectable VAF within 12 months of receiving the first dose of imatinib

  --Abl mutations resistant to imatinib (T315I, F317L/V/C, T315A, V299L, Y253H, E255V/K, F359V/I/C)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imatinib or other agents used in study.
* Concomitant medications that include the following:

  --Participants requiring medications which are inhibitors or inducers of CYP3A4 metabolism, as these may change imatinib plasma levels.
* Uncontrolled intercurrent illness evaluated by history, physical exam, and chemistries or situations that would limit compliance with study requirements, interpretation of results or that could increase risk to the participant
* Participants with the following cardiac conditions: symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Determine the dose of imatinib for dose expansion in participants with pathogenic or likely pathogenic germline RUNX1 mutations during the dose escalation phase | Arm 1 for 1 month and Arm 2 for 3 months
  Safety will be evaluated by the number of DLTs identified at each dose level. The number of DLTs at each dose level will be reported and used to determine the RP2D.
Determine the safety of imatinib in participants with pathogenic or likely pathogenic germline RUNX1 mutations during the dose expansion phase | Arm 1 for 1 month and Arm 2 for 3 months
  Safety will be evaluated by the number of DLTs identified at each dose level.

SECONDARY OUTCOMES:
Pharmacokinetics of imatinib in the RUNX1 population in the dose expansion phase | Measured at baseline (Day 1) and Day 84 for Arm 2
  Change in measurement of drug levels in blood; assessed for potential differences in their study results before and after imatinib administration by an appropriate paired test.
Improvement in platelet dense granule structure by electron microscopy as compared to baseline in the dose expansion phase | Measured at baseline (Day 1- both arms) and Day 84 for Arm 2
  Change in measurement; assessed for potential differences in their study results before and after imatinib administration by an appropriate paired test.
Change in platelet qualitative defects | Measured at baseline (Day 1- both arms) and Day 28 for Arm 1 and Day 84 for Arm 2
  Change in measurement; assessed for potential differences in their study results before and after imatinib administration by an appropriate paired test.
Safety of imatinib in the dose escalation phase | Assessed from Day 1 of study drug through 28 days after the first dose.
  AEs are reported by type and grade, and frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Lea C Cunningham, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.@@@@@@
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers at least 1 year after the completion of the primary endpoint. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active. @@@@@@
Access Criteria: Data from this study may be requested by contacting the PI. Genomic data are made available via dbGaP through requests to the data custodians.@@@@@@

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001542-C.html